CLINICAL TRIAL: NCT03520088
Title: PROSPECTIVE CONTROLLED AND RANDOMIZED STUDY OF THE GENITOURINARY FUNCTION AFTER RECTAL CANCER SURGERY IN RELATION TO THE DISSECTION OF THE INFERIOR MESENTERIC VESSELS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Paula Planelles-Soler (Unknown); Laura Mora-Lopez (Unknown); Naim Hannaoui (Unknown); Sheila Serra-Pla (Unknown); Arturo Dominguez-Garcia (Unknown); Jesus Muñoz-Rodriguez (Unknown); Joan Prats-Lopez (Unknown); Salvador Navarro-Soto (Unknown); Xavier Serra-Aracil (Unknown)
Responsible Party: Principal Investigator, Anna Pallisera-Lloveras, md, PhD, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TAU-RECTALNERV-PRESERV-2018
Record Dates: First submitted 2018-04-03; First posted 2018-05-09 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Sexual dysfunction; Urinary dysfunction; Rectal nerves damage; Total Mesorectal Excision
MeSH Terms: conditions — Rectal Neoplasms; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The analysis of the results will be blind for the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inferior mesenteric Vein dissection (Experimental): To improve and preserve the rectal nerve in the total mesorectal excision, its starts the dissection from the inferior mesenteric vein to the inferior mesenteric artery and through the pelvis
  Interventions: Procedure: Inferior mesenteric Vein dissection
- Inferior mesenteric Artery dissection (Active Comparator): As standard, the dissection starts straight in the inferior mesenteric artery and through the pelvis
  Interventions: Procedure: Inferior mesenteric Artery dissection

INTERVENTIONS:
Procedure: Inferior mesenteric Vein dissection — Dissection of the Inferior mesenteric Vein first, and go down to the Artery during the total mesorectal excision
  Arms: Inferior mesenteric Vein dissection
Procedure: Inferior mesenteric Artery dissection — Dissection of the Inferior mesenteric Artery directly in the total mesorectal excision
  Arms: Inferior mesenteric Artery dissection

SUMMARY:
Purpose: The "Total Mesorectal Excision" (TME) is the standard surgical technique for the treatment of rectal cancer. Up to 50% of sexual dysfunction is described after TME and up to 30% of urinary dysfunction. The main objective of the study is to compare pre- and post-TME sexual dysfunction according to the approach of the inferior mesenteric vessels, directly on the IMA or from the inferior mesenteric vein (IMV) to the IMA.

Methods: Multicenter, prospective, controlled and randomized study of patients with rectal adenocarcinoma with neoadjuvant chemoradiotherapy, who will be randomized into two groups depending on the approach of the inferior mesenteric vessels. The main variable is pre and postoperative sexual dysfunction. The sample to be included will be 90 patients, 45 per group.

DETAILED DESCRIPTION:
Purpose: The "Total Mesorectal Excision" (TME) is the standard surgical technique for the treatment of rectal cancer. Up to 50% of sexual dysfunction is described after TME and up to 30% of urinary dysfunction. Although there are other factors, the main cause of postoperative genitourinary dysfunction is intraoperative injury of the autonomic pelvic nerves. One of the regions with more risk is the Inferior Mesenteric Artery (IMA). The main objective of the study is to compare pre- and post-TME sexual dysfunction according to the approach of the inferior mesenteric vessels, directly on the IMA or from the inferior mesenteric vein (IMV) to the IMA.

Methods: Multicenter, prospective, controlled and randomized study of patients with rectal adenocarcinoma with neoadjuvant chemoradiotherapy, who will be randomized into two groups depending on the approach of the inferior mesenteric vessels. The main variable is pre and postoperative sexual dysfunction. The secondary variables are visualization and preservation of the pelvic autonomic nerves, pre- and postoperative urinary dysfunction, pre and postoperative quality of life. The sample to be included will be 90 patients, 45 per group.

ELIGIBILITY:
Inclusion Criteria:

* Males;
* Age greater (or equal) to 18 years
* Diagnosed of rectal adenocarcinoma at ≤ 15 cm from the anal margin (by rigid rectoscopy)
* Candidate for neoadjuvant (chemoradiotherapy).
* Scheduled laparoscopic radical TME surgery carried out by colorectal surgeons;
* ASA I, II or III;
* Informed consent present.

Exclusion Criteria:

* women
* Under 18 years old;
* Not Candidate for neoadjuvant (chemoradiotherapy);
* Emergency surgery;
* Recurrent neoplasms
* cT4
* Patient with a history of infra-abdominal, or pelvic surgery of the prostate, or radiotherapy prior to the current process;
* Patients with severe sexual dysfunction and neurological alterations before surgery
* Patients with neurogenic bladder before surgery.
* Not to sign the informed consent

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male. The main objective of the study is asses the sexual dysfunction in male
Enrollment: 90 (Estimated)
Dates: Start 2018-09-03 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in sexual dysfunction pre- and post-Total Mesorectal Excision | 1 week before surgery and 12 months post-surgery
  Sexual dysfunction pre- and post-Total Mesorectal Excision by sexual dysfunction scale IIEF-5

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pallisera-Lloveras, MD, PhD, Principal Investigator — Corporacio Parc Tauli. Parc Tauli University Hospital
Locations (1):
- Parc Tauli University Hospital, Sabadell, Barcelona, Spain

REFERENCES:
- [Derived] Pallisera-Lloveras A, Planelles-Soler P, Hannaoui N, Mora-Lopez L, Munoz-Rodriguez J, Serra-Pla S, Dominguez-Garcia A, Prats-Lopez J, Navarro-Soto S, Serra-Aracil X; Tauli-Colorectal Cancer Study Group. Dissection of the inferior mesenteric vein versus of the inferior mesenteric artery for the genitourinary function after laparoscopic approach of rectal cancer surgery: a randomized controlled trial. BMC Urol. 2019 Aug 5;19(1):75. doi: 10.1186/s12894-019-0501-5. PMID 31382934